CLINICAL TRIAL: NCT05903495
Title: A Randomized, Sham-Controlled Trial Investigating Deep Brain Stimulation as a Novel Treatment for Refractory Opioid Use Disorder
Brief Title: Deep Brain Stimulation as a Novel Treatment for Refractory Opioid Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2301715195
Record Dates: First submitted 2023-05-11; First posted 2023-06-15 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-05

CONDITIONS: Opioid-Related Disorders
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: After completion of surgery, participants will be randomly assigned to one of two groups: Group A or Group B. Group A (DBS-ON) will have their stimulator turned on after recovering from surgery. Group B (DBS-OFF) will receive sham stimulation, meaning the stimulator will remain off until Study Week 12 of the outpatient phase, at which time the stimulator will be turned on and left on for the remainder of the study. Group A will continue to receive stimulation and not have the stimulator turned off. participant and assessor will not know which group are assigned to until Study Week 12.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- DBS-ON (Experimental): Titration will be based on stimulation parameters used in previous studies examining the role of DBS of the NAc in the treatment o OCD and depression as well as the parameters utilized in the initial pilot study conducted by the team.
  Interventions: Device: Deep Brain Stimulation
- DBS-OFF (Sham Comparator): For participants randomized to the "DBS-OFF" condition, titration sessions will be conducted identically to the "DBS-ON" arm, the only difference is that no stimulation is delivered and therefore, no actual adjustments made
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — randomized, sham-controlled, partial crossover study investigating DBS, targeting the nucleus accumbens (NAc) and ventral internal capsule (VC), for participants with severe, treatment refractory OUD.

SUMMARY:
The purpose of this clinical study is to investigate the safety, tolerability, and feasibility of Deep Brain Stimulation (DBS) of the nucleus accumbens (NAc) and ventral internal capsule (VC) for participants with treatment refractory opioid use disorder (OUD) who have cognitive, behavioral, and functional disability.

DETAILED DESCRIPTION:
The overarching goal of this study is to evaluate the safety, tolerability, feasibility and impact on outcomes of NAc/VC DBS for treatment refractory OUD. In treatment refractory OUD, innovative approaches and more invasive interventions including DBS are warranted to improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 22-50 years at time of enrollment.
* Fulfills current DSM-5 diagnostic criteria for severe OUD with at least a 5-year history.
* Participants may have comorbid SUD diagnoses at a mild, moderate or severe level, however, OUD must be the primary disorder for which the individual is seeking treatment and the other use disorders must occur in the context of relapse.
* At least one lifetime overdose survival.
* Demonstrated greater than five years of refractory symptoms of OUD.

Exclusion Criteria:

* Diagnosis of acute myocardial infarction or cardiac arrest 1 within the previous 6 months.
* Past or present diagnosis of schizophrenia, psychotic disorder, bipolar disorder, or untreated depression other than one determined to be substance induced.
* Unable to undergo MR-imaging

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as measured by all adverse events related to DBS | Outpatient Week 12
  Incidence of Study-Emergent Adverse Events. The safety/tolerability primary endpoint will be assessed comparing Grade 3 and 4 adverse events between the Active (DBS-ON) and Sham (DBS-OFF) arms throughout Phase IV (Outpatient Week 12). We will also categorize adverse events by organ system and assess relatedness to any aspect of this proof-of-concept study. Statistical tests will be performed at the request of the Data and Safety Monitoring Board (DSMB).
Opioid use assessed via quantitative urine toxicology | Outpatient Week 12
  Opioid use will be evaluated through the use of quantitative urine toxicology using gas chromatography/mass spectrometry. For each subject, quantitative urine toxicology will be collected at baseline (during screening) and during Outpatient Follow-Up Week 4, 8, and 12. The primary outcome comparison between the active and sham arms will be the percentage of participants with undetectable opioid metabolites (assessed via quantitative urine toxicology) throughout the primary Outpatient Week 12 endpoint.

SECONDARY OUTCOMES:
Changes in the Brain Reward Circuitry (FDG PET) | Change from Baseline versus Outpatient Week 12
  Changes in the reward circuitry via evaluating prefrontal cortex glucose metabolism (FDG PET)
Changes in the Brain Reward Circuitry (Fallypride PET) | Change from Baseline versus Outpatient Week 12
  Changes in the reward circuitry via evaluating dopamine in the basal ganglia and NAc (18F-fallypride PET).
Changes in Non-Cue Induced Substance Craving (Visual Analog Scale) | Change from Baseline versus Outpatient Week 12
  Substance craving without cues: Substance craving will be assessed using a visual analog scale (VAS) where participants are asked to rate their craving. Participants will be asked "How much do you crave [insert substance name] right now?".
  Scale: 0 to 10 where 0 = no craving and 10 = maximum craving
Changes in Cue-Induced Substance Craving (Visual Analog Scale) | Change from Baseline versus Outpatient Week 12
  Substance craving with cues (via a cue reactivity task): A set of substance-related stimuli (e.g., photos, computer images) will be presented to the participant. Prior to and immediately after viewing the cues, participants will complete computer-based assessment VAS designed to assess craving. Participants will be asked "How much do you crave [insert substance name] right now?".
  Scale: 0 to 10 where 0 = no craving and 10 = maximum craving
Changes in Mood and Emotional Functioning (Comprehensive Psychopathological Rating Scale) | Change from Baseline versus Outpatient Week 12
  Mood and emotional functioning (depression and anxiety) assessed via the Comprehensive Psychopathological Rating Scale (CPRS)
  Scale: 0 - 108 where 0 = no distress and 108 = severe distress
Changes in Cognitive Functioning (NIH Toolbox Cognition Battery) | Change from Baseline versus Outpatient Week 12
  Cognitive Functioning assessed via NIH Toolbox Cognition Battery (NIHTB)
Changes in Cognitive Functioning (Standard Neuropsychological Battery) | Change from Baseline versus Outpatient Week 12
  Cognitive Functioning assessed via the standard neuropsychological battery (e.g., WAIS-IV)
Changes in Cognitive Functioning (Executive Functioning: Flanker, N-Back, Psychomotor Vigilance, Delayed Discounting) | Change from Baseline versus Outpatient Week 12
  Cognitive Functioning assessed via the experimental measures of executive functioning (e.g., Flanker, N-Back, Psychomotor Vigilance, Delayed Discounting).

CONTACTS AND LOCATIONS:
Overall Officials: James Mahoney, PhD, Study Director — WVU Rockefeller Neuroscience Institute
Locations (1):
- West Virginia University Rockefeller Neuroscience Institute, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No